CLINICAL TRIAL: NCT00783939
Title: Safety Dermatological Evaluation: Vaginal Mucous Irritation - Product Tested: Dermacyd PH_DETINBACK Tangerine Mix (Lactic Acid).
Brief Title: Dermacyd PH_DETINBACK Tangerine Mix (Lactic Acid) - Safety.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04307
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Lactic Acid (Dermacyd PH_DETINBACK Tangerine Mix)
  Interventions: Drug: Lactic Acid

INTERVENTIONS:
Drug: Lactic Acid — Lactic Acid (Dermacyd PH_DETINBACK Tangerine Mix)

SUMMARY:
The purpose of this study is to prove the safety in normal conditions of useof the product Dermacyd PH_DETINBACK Tangerine Mix (Lactic Acid).

ELIGIBILITY:
Inclusion criteria:

* Age between 10 and 20 years old;
* Integral skin test in the region;
* Use of cosmetic product of the same category;
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time;

Exclusion criteria:

* Lactation or gestational risk or gestation;
* Use of Anti-inflammatory, immunosuppression or antihistaminic drugs;
* Atopic antecedent or allergic to cosmetic product;
* Active cutaneous disease in the evaluation area;
* Diseases which cause immunology decrease, such as diabetes and HIV;
* Endocrinal pathologies;
* Intense solar exposure 15 days before the evaluation;
* Treatment until four months before the selection;

The above information is not intended to contain all considerations relevant to a patient¿s potential participation in a clinical trial.

Ages: 10 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The absence of irritation and the good acceptability will be evaluated using one specific scale which describes the intensity of the reaction. | From the treatment start to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil